CLINICAL TRIAL: NCT07115693
Title: Comparison of Upper Extremity Resistance Exercises as Synchronous Tele and Home Programs in Paraplegic Patients: a Randomized, Controlled, Double-blind Study
Brief Title: Synchronous Tele-Resistance Training to Improve Upper Extremity Function in Patients With Spinal Cord Injury
Acronym: TELERES-SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacer Önen Tekin (Other)
Responsible Party: Sponsor-Investigator, Hacer Önen Tekin, investigator, Istinye University
Organization: Istinye University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IST-FTR-TELERES-SCI-2025
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Telerehabilitation with Resistance Exercises (Experimental): Participants received live, video-based supervised resistance training 3x/week for 6 weeks.
  Interventions: Behavioral: Telerehabilitation-Based Resistance Exercise Program
- Home-Based Exercise Program (Active Comparator): Participants followed an unsupervised exercise program at home for 6 weeks.
  Interventions: Behavioral: Home Exercise Program

INTERVENTIONS:
Behavioral: Telerehabilitation-Based Resistance Exercise Program — Participants received synchronous telerehabilitation sessions three times per week for six weeks. Each session lasted 45 minutes and included supervised resistance exercises for upper extremity muscle groups. Exercise bands were chosen based on baseline strength. Pulse oximeters were used to monitor heart rate and oxygen saturation.
  Arms: Synchronous Telerehabilitation with Resistance Exercises
Behavioral: Home Exercise Program — Participants were given a home-based, unsupervised exercise program to follow three times per week for six weeks. The exercises were taught at the beginning, and adherence was monitored using a physical activity diary. No tele-supervision was provided.
  Arms: Home-Based Exercise Program

SUMMARY:
This study investigated the effects of resistive exercises applied with synchronized telerehabilitation on upper extremity functions in patients with SCI who use wheelchairs. A randomized controlled trial included 21 patients with SCI between the ages of between18 and 60. Participants were divided into two groups: the Study Group (n=11) and the Control Group (n=10). Participants in the study group applied resistive exercise with a synchronized telerehabilitation method, while participants in the control group applied a home exercise program. The upper extremity muscle strength of the participants was evaluated with hand-held dynamometer before and after the treatment, physical performance with a 20-meter push test, and physical activity level with Physical Activity Scale for Disabled Individuals.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years
* Diagnosed with spinal cord injury classified as ASIA A, B, or C
* Cooperative and able to follow verbal instructions
* Has access to online communication devices
* Partially or fully dependent on a wheelchair
* Sufficient upper extremity strength to operate a wheelchair
* Has not undergone surgery in the past 6 months
* Willing to participate and provided informed consent

Exclusion Criteria:

* Unwilling or unmotivated to participate
* Presence of a progressive disease
* Fully bedridden
* Significant cognitive impairment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change in upper extremity muscle strength measured by hand-held dynamometer | Baseline and after 6 weeks of intervention
  Muscle strength of the shoulder flexors, extensors, abductors, and wrist flexors and extensors will be measured bilaterally using a hand-held dynamometer. The outcome is reported in Newtons (N).

CONTACTS AND LOCATIONS:
Locations (1):
- Turkish Spinal Cord Paralytics Association at Hüsnü Ayık Special Care Center, Diyarbakır, Kayapınar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided